CLINICAL TRIAL: NCT03398187
Title: Cardiac Catheterization in the Management of Pediatric Cardiac Patients at Assiut University Children Hospital ( A Descriptive Study)
Brief Title: Cardiac Catheterization in the Management of Pediatric Cardiac Patients at A.U.C.H.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen Ahmed Mahmoud Sayed, Doctor, Assiut University
Other Study IDs: Cardiac Cath. at A.U.C.H.
Record Dates: First submitted 2017-12-12; First posted 2018-01-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Cardiac Catheterization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiac catheterization — diagnostic and interventional cardiac catheterization

SUMMARY:
The aim of this study is to find out and record the indications for diagnostic catheterization as well as for interventional cardiac catheterization in A.U.C.H , and record the outcome in these cases.

DETAILED DESCRIPTION:
Cardiac catheterization is of two types:

diagnostic and interventional . There has been recent advances in these procedures.There is an over 10y experience at the pediatric cardiology unit in assiut University Children Hospital ( A.U.C.H ) catheterization department. The procedure usually follows other investigations used for evaluation of the pediatric cardiac patients e.g. chest X-ray , ECG and echocardiography.

The role of cardiac catheterization may be in the diagnosis of congenital cardiac anomalies as well as in the follow up of repair of some cardiac anomalies . On the other hand, the indications for interventional cardiac catheterization may be repair of Atrial septal defect, Transposition of great arteries palliation with balloon septostomy ,blood vessel dilatation e.g. aortic stenosis and coarctation of the aorta . In addition Patent ductus arteriosus closure and others may be done by the interventional cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

-all cases admitted for cardiac catheterization for diagnosis or intervention at Assiut University Children Hospital

Exclusion Criteria:

* cases not admitted for diagnostic or interventional cardiac catheterization

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all cases admitted for cardiac catheterization for diagnosis or intervention at Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
procedure time | duration of the cardiac catheterization procedure (1-4 hours depending on complexity of case)
  duration of the cardiac catheterization procedure (1-4 hours depending on complexity of case|)

REFERENCES:
- See also: pediatric cardiac catheterization databases — https://jhu.pure.elsevier.com/en/publications/pediatric-cardiac-catheterization-databases-4